CLINICAL TRIAL: NCT04106232
Title: MIcrobiome Analysis of Chronically Constipated Versus Non-constipated Populations for Detection of Novel Molecular Entities With Therapeutic Potential
Brief Title: Microbiome Analysis of Constipated Versus Non-constipation Patients
Status: Completed | Type: Observational
Sponsor: HyGIeaCare, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HGP-0008
Record Dates: First submitted 2019-09-20; First posted 2019-09-26 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-11

CONDITIONS: Rome IV Functional Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Overall, we expect to enroll 20 subjects. Each volunteer or patient will provide a traditional stool sample ("spot sample"), collected in their home. During the HyGIeaCare prep, we will collect up to 3 samples from each patient (unless we will need an "initial" one from the constipated population).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No change in procedure except for specimen collection throughout procedure — Stool specimens will be taken before and during the HyGIeaCare procedure. Microbiome comparisons will be made across all specimens

SUMMARY:
This study intends to evaluate the microbiome of chronically constipated patients as compared to those with a non-constipated gastrointestinal system.

DETAILED DESCRIPTION:
Biogeographically accurate microbiome sampling using the HyGIeaCare platform and an evolutionary biology informed learning platform will allow an improved discovery of bacterially derived novel molecular entities with therapeutic potential for chronic constipation. This approach intends to enhance our ability to understand the gut microbiome and use it towards developing therapeutic solutions, in comparison to traditional collection methods and taxonomic-based data analysis approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age is between 18 and 80 years old.
2. For the healthy population - Indication for age-appropriate colorectal cancer screening colonoscopy
3. Adequate capacity to consent to study
4. Patient does not have any known health issues, except for chronic constipation for the "chronic constipation" population.
5. Patient has not taken antibiotics within the last three (3) months.
6. For chronically constipated patients - >3 months of symptomatic constipation with first onset of constipation more than 6 months ago.

For chronically constipated patients - Diagnosis of functional constipation by Modified Rome IV Diagnostic Criteria.

Exclusion Criteria:

1. Patient has functional bowel disorders characterized by alternating bowel habits (diarrhea/constipation).
2. Patient has any other condition that, in the opinion of the investigator, may adversely affect the compliance or safety of the patient or would limit the patient's ability to complete the study.
3. Current, or recent (within three months) antibiotic usage

   Patient has any of the contraindications listed below:
4. Cardiac: Congestive heart failure (NYHA class III or IV or EF <50%)
5. GI: Intestinal perforation, carcinoma of the rectum, fissures or fistula, severe hemorrhoids, abdominal hernia, recent colon or rectal surgery, or abdominal surgery
6. GU: Renal insufficiency (CC < 60 ml/min/173m2), cirrhosis with ascites
7. Abdominal surgery within the last 6 months
8. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and chronically constipated patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Identify the presence of microbial substances within stool samples taken from different locations along the colon | 12 months
  Finding novel molecular entities with therapeutic potential for chronic constipation using the unique HyGIeaCare approach for constipation relief and collection of fecal material for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: David A Johnson, MD, Principal Investigator — Eastern Virginia Medical School
Locations (3):
- United States (3):
  - Hygieacare Center - Flowood, Flowood, Mississippi
  - Hygieacare - Norwood, Cincinnati, Ohio
  - HyGIeaCare Center, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
Outcomes will be used internally for future studies.